CLINICAL TRIAL: NCT05359510
Title: The Use of Different Types of Mesh at Different Sites in the Prevention of Incisional Hernia After Various Abdominal Incision Versus Primary Abdominal Suturing.
Brief Title: The Use of Different Types of Mesh for Prevention of Incisional Hernia Versus Primary Abdominal Suturing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kerolos Samer Shafik, Assistant Lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I H repair by mesh
Record Dates: First submitted 2022-04-25; First posted 2022-05-04 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Incisional Hernia
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient with various abdominal incisions to be operated (Experimental): patients with various abdominal incisions for closure either by primary suturing or by mesh
  Interventions: Procedure: prophylactic mesh repair at different sites for prevention of incisional hernia after various abdominal incision versus primary abdominal suturing

INTERVENTIONS:
Procedure: prophylactic mesh repair at different sites for prevention of incisional hernia after various abdominal incision versus primary abdominal suturing — before closure of the abdominal layers prophylactic mesh will be used for prevention of incisional hernia. another patient with abdominal incision , primary closure of abdominal layer will occur.
  Other Names: closure of various abdominal incision by different types of prophylactic mesh at different sites for prevention of incisional hernia versus primary abdominal closure

SUMMARY:
The use of different types of mesh at different sites in prevention of incisional hernia after various abdominal incision versus primary abdominal suturing.

DETAILED DESCRIPTION:
The burden of incisional hernia after abdominal exploration has raised the question if a prophylactic mesh placement during abdominal wall closure is of benefit.

The reported rate of incisional hernia after abdominal incisions varies from 4.2% up to a calculated risk of 73%. The impact on quality of life and annual health care costs has motivated various groups to research ways to decrease the rate of incisional hernia by optimizing the technique of abdominal wall closure.

One of the crucial risk factors of the genesis of incisional hernias is the malfunction of collagen synthesis. Other main risk factors are found to be obesity, steroid therapy, malnutrition, nicotine abuse, and other connective tissue diseases.

Since German physician Theodor Billroth's first suggested use of prosthetic material to close the hernia defect in 1890, continued interest lead to the development of a variety of surgical meshes and techniques for suture and mesh reinforcement to prevent incisional hernia . Overtime, RCTs have demonstrated the effectiveness of the use of prophylactic mesh in the prevention of incisional hernia. While surgeons world over use different techniques of positioning mesh in the prophylactic mesh repair (PMR) such as the Onlay, Sublay and Intraperitoneal positions, which can be associated with a high incidence of complications such as the postoperative seroma.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* patient age: ≥ 18 years
* patients undergoing elective or urgent open abdominal surgical procedure regardless of benign or malignant disease

Exclusion Criteria:

* age <18 years
* navel site infection
* pregnancy
* expected survival <12 month
* previous intra abdominal mesh placement

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
early wound complications | 1 month
  wound infection (with or without removal of the mesh) ,wound necrosis , wound hematoma
late wound complications | 1 month
  post operative incisional hernia, wound infection (with or without removal of the mesh) wound necrosis wound hematoma.

SECONDARY OUTCOMES:
complication rate | intraoperative complications will be recorded immediately after finishing the operation
  major bleeding bowel injury
incidence of incisional hernia | 12 month
  the incidence of incisional hernia, either symptomatic or asymptomatic in the mesh and suture-only groups.

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Abdel Aziz, Study Chair — general surgery Assiut universitiy
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
age ,sex ,clinical diagnosis
Supporting Information: Study Protocol, SAP
Time Frame: 3 years
Access Criteria: age ,sex, clinical diagnosis